CLINICAL TRIAL: NCT04768764
Title: Comparison Of Femoral Block And Middle Adductor Canal Block In Patients With Knee Arthroplasty In Terms Of Postoperative Pain Control And Early Mobilization
Brief Title: Comparison Of Femoral Block And Middle Adductor Canal Block In Patients With Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Elif Göktaş, Anesthesiology Resident, Bozyaka Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: elifgoktas
Record Dates: First submitted 2021-02-22; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative; Anesthesia and Analgesia; Anesthesia, Conduction; Nerve Block
Keywords: femoral nerve block; adductor block; knee arthroplasty
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Anesthesia, Conduction; Bupivacaine; Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: There are two groups: the first group is adductor block and the second group is femoral block.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Middle Adductor Canal Block (Active Comparator): Ultrasound Guided Middle Adductor Canal Block:
  20 ml Bupivacaine 0.25% Injectable Solution will be administered for middle adductor canal block.
  10 ml %0,5 Bupivacaine will be diluted with 10 ml saline solution.
  Interventions: Procedure: Ultrasound Guided Middle Adductor Canal Block; Drug: Bupivacain; Procedure: Spinal Anesthesia
- Group 2 Femoral Nerve Block. (Active Comparator): Ultrasound Guided Femoral Nerve Block:
  20 ml Bupivacaine 0.25% Injectable Solution will be administered for femoral nerve block.
  10 ml %0,5 Bupivacaine will be diluted with 10 ml saline solution.
  Interventions: Procedure: Ultrasound Guided Femoral Nerve Block.; Drug: Bupivacain; Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: Ultrasound Guided Middle Adductor Canal Block — Middle adductor canal block will be applied post-operatively with guidance of USG.
  Drug:Bupivacaine 0.25% Injectable Solution
  Other Names: Regional Anesthesia
  Arms: Group 1 Middle Adductor Canal Block
Procedure: Ultrasound Guided Femoral Nerve Block. — Femoral nerve block will be applied post-operatively with guidance of USG. Drug:Bupivacaine 0.25% Injectable Solution
  Other Names: Regional Anesthesia
  Arms: Group 2 Femoral Nerve Block.
Drug: Bupivacain — 10 ml %0,5 Bupivacaine will be diluted with 10 ml saline solution. Bupivacaine 0.25% Injectable Solution
  Other Names: Marcain
Procedure: Spinal Anesthesia — Patients will be placed in the lateral decubitus position.Subarachnoid space will be entered through the most suitable intervertebral space.Bupivacaine 0.5% Heavy will be given in the appropriate dose.

SUMMARY:
Femoral and adductor nerve blocks with ultrasonography(USG) guidance are used effectively and efficiently in post-operative pain management in lower extremity surgical procedures. However, the superiority of these two blocks to each other is still controversial. In this prospective, randomized, double-blind study, patients who underwent elective unilateral knee arthroplasty under spinal anesthesia, will be performed postoperative femoral block or middle adductor canal block with the guidance of USG.Patients who underwent spinal anesthesia and needed sedoanalgesia and who had to switch to general anesthesia will be excluded from the study. The patients will be divided into two groups by simple randomization. Since a total of 52 patients should be included in the study as a result of the power analysis (G-power 3.1); It is planned to take approximately 26 patients for each group.The anesthesiologist, who follows the pain control and mobilization after the block, will not know which study group the patient is in. The blocks will be performed behind the cover while the patient is under spinal anesthesia (Thus, the point of application of the block will not be noticed). In this way, the patient and the anesthesiologist who follows the parameters after the block will be blind to patient's arm. In the first group, 0.25% 20 ml of local anesthetic and middle adductor canal block, in the second group 0.25% 20 ml of local anesthetic and femoral nerve block will be applied We will compare these two blocks in terms of early mobilization, postoperative pain control, motor, and sensory block.

DETAILED DESCRIPTION:
All patients scheduled for total knee arthroplasty will be evaluated before the operation. Eligible patients will be informed about the study and "Numeric Rating Scale" for pain evaluation. Then, patients will be asked for informed consent. After approval from the local research ethics committee, first patient will be recruited for study and patient's group will be determined by dice roll. Patients who are scheduled for primary total knee arthroplasty under spinal anesthesia with a planned sensory block level between T4 and T7 dermatomes, will be recruited and assigned to a group.Femoral block or middle adductor canal block will be applied to the patients.

Group1 (Group 1 Middle Adductor Canal Block) patients will be administered middle adductor canal block with 20 ml 0.25% Bupivacaine by an experienced anesthesiologist.

Group2 (Femoral Nerve Block) patients will be administered femoral block with 20 ml 0.25% Bupivacaine by an experienced anesthesiologist.

The selected block will be applied with USG behind the curtain after the operation.Patients will be taken to the postoperative recovery unit.Patients will be followed-up in post-anesthesia care unit and in the ward for 48 hours. Post-operatively, patients will receive 1mg/kg Tramadol when Numeric Rating Scale(NRS) > 3.The duration of the sensory and motor block and the mobilization of the patients will be recorded and compared.

0,2,4,6,8,12,24 of the patient pain scores at hour and 6 months, presence of sensory block and motor block, pain score when the patient is mobilized will be recorded.In addition, operation time, complications related to block, mobilization time, discharge day, and opioid need will be recorded.It will be recorded at what time the first opioid dose was administered after the block.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2-3 patients who will undergo unilateral elective primary total knee prosthesis surgery with consent for the study
* Patients whose operation has been successfully completed with spinal anesthesia

Exclusion Criteria:

* Refusal of the patient to work
* Patients under 18 years of age
* Patients who have undergone an anesthesia technique other than spinal anesthesia for any reason (general anesthesia, sedoanelgesia, laryngeal mask application, etc.)
* Those with known local anesthetic allergies
* Body mass index> 35 patient groups
* Skin infection at the injection site
* Coagulopathy and use of anticoagulant therapy
* Uncontrolled diabetic patients
* Uncooperative patient
* Physiological and emotional lability
* Prolonged surgical intervention
* Patient with limitation of mobilization and movement before the operation, other than the operation reason

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-04-16 (Estimated); Primary Completion 2021-10-16 (Estimated); Study Completion 2022-04-16 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 0th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 0th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 2nd hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 2nd hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 4th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 4th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 6th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 6th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 8th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 8th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 12th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 12th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 24th hour postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 24th hour postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 6 months postoperatively
  Pain scores will be recorded as reported by the patient according to NRS
Post-operative pain assessed by Numeric Rating Scale(NRS) | At 6 months postoperatively
  Pain scores will be recorded as reported by the patient while knee flexion according to NRS
Ambulation time | 48 hours postoperatively
  First time a patients can walk around independently
NRS at Ambulation | 48 hours postoperatively
  NRS when first time a patients can walk around independently

SECONDARY OUTCOMES:
Time of First Rescue Opioid | 48 hours postoperatively
  When patient's pain score(NRS) is 3 or more.
Time of Return of Sensory Block | 24 hours postoperatively
  Examined with Prick Test
Time of Return of Motor Block | 24 hours postoperatively
  Examined with Examined with Holmenn Skalası

CONTACTS AND LOCATIONS:
Overall Officials: Zeki Tuncel Tekgül, Study Director — İzmir Bozyaka Training and Research Hospital
Locations (1):
- İzmir Bozyaka Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No